CLINICAL TRIAL: NCT03111797
Title: Robot-assisted Lobectomy Versus Video-assisted Lobectomy : a Prospective Observational Study
Brief Title: Robot-assisted Lobectomy Versus Video-assisted Lobectomy
Status: Completed | Type: Observational
Sponsor: Hospital Nord (Other)
Collaborators: Gary DUCLOS (Medical Doctor, investigator) (Unknown)
Responsible Party: Principal Investigator, marc LEONE, Study Director, Clinical professor, Hospital Nord
Other Study IDs: darnord2017-02
Record Dates: First submitted 2017-04-08; First posted 2017-04-13 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Robotic Surgical Procedures; Pneumonectomy; Status; Anesthesia and Analgesia; Cardiac Output
MeSH Terms: conditions — Agnosia | interventions — Morphine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- video-assisted lobectomy group: patients operated of lung lobectomy for an early stage cancer using a video-assisted surgical procedure
  Interventions: Drug: Morphine; Other: Cardiac output measure
- robot-assisted lobectomy group: patients operated of lung lobectomy for an early stage cancer using a robot-assisted surgical procedure
  Interventions: Drug: Morphine; Other: Cardiac output measure

INTERVENTIONS:
Drug: Morphine — we observe the self-patient controlled morphine consumption during the first 48h after surgery
Other: Cardiac output measure — we observe the cardiac output during surgical procedure using a non-invasive cardiac output monitoring device (ClearSight from Edwards lifescience laboratory )

SUMMARY:
This prospective and observational cohort studies the morphine consumption difference during the first 48 hours after a lung lobectomy between patients operated with a robot assisted or a video-assisted technique for a lung cancer lobectomy.

Second outcome was to search eventual cardiac output difference during the surgery in 100 patients (50 in each group) using a non invasive monitoring device of cardiac output

All patients operated between january 2016 and March 2017 for a lung cancer lobectomy were included.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers
* Mono lobectomy of lung for early stage cancer (T2Nx and earlier)
* Video or robot assisted procedure

Exclusion Criteria:

* Advanced stage of cancer (T3Nx and greater)
* Need of thoracotomy conversion during procedure
* Morphine intolerance or addiction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients needing a lung lobectomy surgery for an early stage cancer in our center during the period of inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | 48 hours after surgery
  morphine consumption for each patient using a self patient - controled morphine pump

SECONDARY OUTCOMES:
cardiac output | during 30 minutes after incision and optic introduction
  continuous cardiac output during surgery procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Departement anesthesie reanimation hopital nord, Marseille, France

IPD SHARING:
Plan to Share IPD: No